CLINICAL TRIAL: NCT01424332
Title: A Randomized, Open Label, Three-way Crossover Study to Evaluate the Pharmacodynamic Interactions Between Darexaban (YM150)/Darexaban Glucuronide (YM-222714) and Acetyl Salicylic Acid (ASA) in Healthy Male Subjects
Brief Title: To Evaluate Whether Acetyl Salicylic Acid (Aspirin) and Darexaban (YM150) Interact in Their Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 150-CL-034; 2007-002194-31 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Pharmacodynamic and Pharmacokinetic Interaction; Healthy Subjects
Keywords: Pharmacodynamics; pharmacokinetics; darexaban; Acetyl Salicylic Acid; darexaban glucuronide; YM150; YM-222714; Phase 1
MeSH Terms: interventions — darexaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment arm 1 (Experimental): darexaban, wash-out, ASA, wash-out, darexaban plus ASA
  Interventions: Drug: Darexaban; Drug: Acetyl Salicylic Acid (ASA)
- Treatment arm 2 (Experimental): darexaban, wash-out, darexaban plus ASA, wash-out, ASA
  Interventions: Drug: Darexaban; Drug: Acetyl Salicylic Acid (ASA)
- Treatment arm 3 (Experimental): ASA, wash-out, darexaban, wash-out, darexaban plus ASA
  Interventions: Drug: Darexaban; Drug: Acetyl Salicylic Acid (ASA)
- Treatment arm 4 (Experimental): ASA, wash-out, darexaban plus ASA, wash-out, darexaban
  Interventions: Drug: Darexaban; Drug: Acetyl Salicylic Acid (ASA)
- Treatment arm 5 (Experimental): darexaban plus ASA, wash-out, darexaban, wash-out, ASA
  Interventions: Drug: Darexaban; Drug: Acetyl Salicylic Acid (ASA)
- Treatment arm 6 (Experimental): darexaban plus ASA, wash-out, ASA, wash-out, darexaban
  Interventions: Drug: Darexaban; Drug: Acetyl Salicylic Acid (ASA)

INTERVENTIONS:
Drug: Darexaban — oral
  Other Names: YM150
Drug: Acetyl Salicylic Acid (ASA) — oral
  Other Names: Aspirin

SUMMARY:
The primary objective of this study is to evaluate whether ASA and darexaban which have different effects on blood coagulation influence each other in their effects. Also it will be investigated whether the blood levels of either drug are influenced by the presence of the other drug. In addition, the safety and tolerability of each drug and the combination of the drugs will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5-30.0 kg/m2
* Male subjects must be non-fertile, i.e. surgically sterilized or must practice an adequate contraceptive method to prevent pregnancies

Exclusion Criteria:

* Known or suspected hypersensitivity to darexaban or ASA or any components of the formulation used
* Any of the liver function tests (i.e. ALT, AST and bilirubin) above the upper limit of normal at repeated measures
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Use of any prescribed or OTC (over-the-counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampicin) in the 3 months prior to admission to the Clinical Unit
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse, or smoking of more than 10 cigarettes (or equivalent) or more than 21 units (210 g) of alcohol per week within the 3 months prior to study
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Composite assessment of pharmacodynamics of darexaban and darexaban glucuronide | Baseline and after six days of dosing of darexaban, ASA, or a combination of the two
  Assessment includes skin bleeding time, factor Xa, platelet aggregation, thromboxane B2 synthesis, PT & aPTT

SECONDARY OUTCOMES:
Pharmacokinetics of darexaban and darexaban glucuronide assessed by plasma concentration | Plasma samples are taken until 24 hours after six days of dosing of darexaban, or the combination with ASA
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG), clinical safety laboratory and adverse events | 6 days for each of the 3 treatment periods
Pharmacokinetics of ASA assessed by plasma concentration | Plasma samples are taken until 2 hours after six days of dosing of ASA, or the combination with darexaban

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.; Principal Investigator, Principal Investigator — SGS Aster, Paris, France
Locations (1):
- SGS Aster, Paris, France